CLINICAL TRIAL: NCT00094887
Title: A Prospective, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of Nitric Oxide for Inhalation in the Acute Treatment of Sickle Cell Pain Crisis
Brief Title: Nitric Oxide Inhalation to Treat Sickle Cell Pain Crises
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INOT 36; 05-H-0019 (Registry Identifier: NIH); NCT00652535 (obsolete NCT alias)
Record Dates: First submitted 2004-10-28; First posted 2004-10-28 (Estimated); Results first posted 2010-04-23 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2017-10

CONDITIONS: Anemia, Sickle Cell
Keywords: Blood Flow; Nitric Oxide; Pain Crisis; Sickle Cell Anemia; Vaso-Occlusive Crisis; Sickle Cell Disease; SCD
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Nitric Oxide; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide (Experimental): Participants receive Inhaled nitric oxide (INO)
  Interventions: Drug: Nitric Oxide
- Placebo (Placebo Comparator): Participants receive Nitrogen gas
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric Oxide — Nitric oxide will be delivered for 4 hours at 80 ppm through a face mask. The dose will then be reduced to 40 ppm for 4 hours. After a total of 8 hours of treatment through face mask, the patient will get 6 mL/puls/breath of NO at 800 ppm or 3 m//pulse/breath, depending on patient weight.
  Other Names: INOmax
  Arms: Inhaled Nitric Oxide
Drug: Placebo — Nitrogen gas will be delivered in the same manor as the experimental drug.
  Arms: Placebo

SUMMARY:
This study will examine whether nitric oxide (NO) gas can reduce the time it takes for pain to go away in patients who are in sickle cell crisis. NO is important in regulating blood vessel dilation, and consequently, blood flow. The gas is continuously produced by cells that line the blood vessels. It is also transported from the lungs by hemoglobin in red blood cells.

Patients 10 years of age or older with sickle cell disease (known SS, S-beta-thalassemia or other blood problems causing sickle cell disease) may be eligible for this study. Patients whose disease is due to hemoglobin (Hgb) SC are excluded. Candidates are screened with blood tests and a chest x-ray to look at the lungs and heart.

Participants are admitted to the hospital in a pain crisis. They are evaluated and then randomly assigned to receive one of two treatments: 1) standard treatment plus NO, or 2) standard treatment plus placebo. The placebo used in this study is nitrogen, a gas that makes up most of the air we breathe and is not known to help in sickle cell disease.

For the first 8 hours of the study, patients receive placebo or NO through a facemask. The mask may be taken off for 5 minutes every hour and for not more than 20 minutes to eat a meal. After the first 8 hours, the gas is delivered through a nasal cannula (small plastic tubing that rests under the nose) that may be taken off only while showering or using the restroom. Patients are questioned about the severity of their pain when they start the study and then every few hours while they are in the hospital. Their vital signs (temperature, breathing rate, and blood pressure) and medicines are checked. Patients will breathe the gas for a maximum of 3 days, but will stay hospitalized until the patient feels well enough to go home. Patients are followed up about 1 month after starting the study by a return visit to the hospital or by a phone call.

DETAILED DESCRIPTION:
The object of this study is to determine the safety and efficacy of nitric oxide for inhalation in the treatment of vaso-occlusive pain crisis (VOC) in patients with sickle cell disease. The study population will include patients with sickle cell disease (SS, S-beta-Thalassemia) presenting with vaso-occlusive pain crisis. Patients will be administered either placebo or inhaled nitric oxide to see if the experimental agent, inhaled nitric oxide, can reduce the time it takes for resolution of the vaso-occlusive crisis.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following inclusion criteria during the screening process in order to participate in the study:

* Patient must have a diagnosis of SCD (known SS, S-Beta-thalassemia or other hemoglobinopathies causing sickle cell disease). Patients with disease due to Hgb SC are not permitted.
* Must present to the ED/EC or other appropriate unit in VOC.
* Greater than or equal to 10 years old.
* Written informed consent/assent has been obtained.

Exclusion Criteria:

Subjects meeting any of the following criteria during baseline evaluation will be excluded from entry into the study:

* Exposure to therapeutic nitric oxide within the past 12 hours.
* Patient has received sildenafil or other phosphodiesterase 5 inhibitors, therapeutic L-arginine, nitroprusside or nitroglycerine within the past 12 hours.
* Patient has received previous ED/EC or other appropriate unit treatment for a vaso-occlusive crisis less than 48 hours or hospitalization less than 14 days ago (patients transferred directly from another ED or clinic may be enrolled).
* Patient has visited the ED/EC or other appropriate unit greater than 10 times in the past year having a vaso-occlusive crisis.
* Patients presenting with clinically diagnosed bacterial infection (e.g., osteomyelitis, pneumonia, sepsis or meningitis).
* Patients who are currently enrolled in any other investigational drug study except for hydroxyurea studies.
* Pregnant women (urine HCG + )/ nursing mothers.
* Patients who have received an exchange transfusion (not simple transfusion) in the last 30 days or are on a chronic simple or exchange transfusion program.
* Suspected splenic sequestration.
* Acute chest syndrome or pneumonia: Abnormal new pulmonary infiltrate (alveolar infiltration and not atelectasis) and one or more pulmonary signs and/or symptoms (fever, rales, wheezing, cough, shortness of breath, retractions).
* Previous participation in this study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Baldassarre, MD, Study Director — Mallinckrodt
Locations (11):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - Children's Hospital Oakland, Oakland, California
  - Colorado Sickle Cell Treatement and Research Center, Aurora, Colorado
  - Howard University Hospital, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Childrens Hospital, Boston, Boston, Massachusetts
  - Case Western Reserve University Hospital, Cleveland, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Childrens Hospital, Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanders DY, Severance HW, Pollack CV Jr. Sickle cell vaso-occlusive pain crisis in adults: alternative strategies for management in the emergency department. South Med J. 1992 Aug;85(8):808-11. doi: 10.1097/00007611-199208000-00005. PMID 1302470
- [Derived] Gladwin MT, Kato GJ, Weiner D, Onyekwere OC, Dampier C, Hsu L, Hagar RW, Howard T, Nuss R, Okam MM, Tremonti CK, Berman B, Villella A, Krishnamurti L, Lanzkron S, Castro O, Gordeuk VR, Coles WA, Peters-Lawrence M, Nichols J, Hall MK, Hildesheim M, Blackwelder WC, Baldassarre J, Casella JF; DeNOVO Investigators. Nitric oxide for inhalation in the acute treatment of sickle cell pain crisis: a randomized controlled trial. JAMA. 2011 Mar 2;305(9):893-902. doi: 10.1001/jama.2011.235. PMID 21364138
- See also: NIH Clinical Center Detailed Web Page — https://www.ncbi.nlm.nih.gov/m/pubmed/1302470/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 11 study centers in the United States
Pre-assignment Details: Of the 150 participants recruited, 150 were randomized (1:1) into treatment groups.
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide | Placebo
Started | 75 | 75
Safety Population | 75 | 75
Intent to Treat Population | 75 | 75
Per Protocol Analysis Set | 71 | 71
Primary Efficacy Population | 65 | 64
Completed | 71 | 71
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Inhaled Nitric Oxide: Inhaled Nitric Oxide INO
- Placebo: Nitrogen gas
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Placebo | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Customized [Number; unit: participants]
  < 16 years | 12 | 14 | 26
  >=16 years | 63 | 61 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (11.06) | 26.0 (10.49) | 26.3 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 37 | 38 | 75
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Time to Vaso-occlusive Pain Crisis (VOC) Resolution
Description: VOC resolution was defined by all of the following conditions:
  * Pain relief - Visual Analog Scale (VAS) pain scores of 6 or less, (6 as worst and 0 as best)
  * Freedom from parenteral narcotic use,
  * Ability to walk unless the subject was not able to walk for any reason other than acute VOC prior to the onset of crisis,
  * Subject and/or family's belief that the painful crisis could be managed at home with or without oral analgesic use, and the physician concurred with that assessment.
Time Frame: within 30 days
Population: Primary efficacy analysis set, defined as intent to treat population with VOC resolution
Measure: Median (Full Range); unit: Hours
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 65 | 64
Hours | 61.83 [9.93 to 412.17] | 55.16 [8.00 to 233.00]
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide vs Placebo; Test type: Other; p = 0.8085, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Length of Hospitalization
Description: Length of hospitalization is defined as the length of time from admission to discharge order
Time Frame: within 40 days
Population: Intention to treat
Measure: Median (Full Range); unit: Days
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 75 | 75
Days | 4.06 [0.76 to 21.35] | 3.11 [0.05 to 39.02]

3. Secondary Outcome: Number of Participants Discharged to Home Within the First 24 Hours
Time Frame: within 24 hours
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 75 | 75
Participants | 5 | 7

4. Secondary Outcome: Total Dose of Opioids Received
Description: The total dose (mg) of opioid medications received during the trial
Time Frame: within 8 hours and within 40 days
Population: Intention to treat
Measure: Median (Full Range); unit: mg
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 75 | 75
mg
  within 8 hours | 16.25 [0.00 to 196.50] | 17.25 [0.00 to 440.00]
  within 40 days | 153.75 [1.60 to 3117.80] | 211.37 [2.00 to 7506.2]

5. Secondary Outcome: Number of Participants With Acute Chest Syndrome/Pneumonia Requiring Blood Transfusion
Description: Number of participants who required a blood transfusion before discharge because of acute chest syndrome/pneumonia
Time Frame: within 40 days
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 75 | 75
Participants | 8 | 7

6. Secondary Outcome: Number of Participants Readmitted to Hospital Within 30 Days After Discharge
Description: The number of participants readmitted to the hospital for any reason within 30 days after discharge
Time Frame: during first 24 hours and during 30 day follow-up
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 75 | 75
Participants
  during first 24 hours | 0 | 0
  during 30-day follow-up | 9 | 17

ADVERSE EVENTS:
Description: 75 subjects were assigned to treatment with iNO and 75 subjects were assigned to treatment with placebo; all subjects were included in the ITT and Safety Populations. 142 subjects completed the study according to the protocol and 8 subjects (4 in each treatment group) did not complete the study according to protocol.
Arm/Group | Inhaled Nitric Oxide | Placebo
Serious Adverse Events (participants affected / at risk) | 7/75 | 6/75
Other Adverse Events (participants affected / at risk) | 35/75 | 33/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (N=75) | Placebo (N=75)
Acute Chest Syndrome (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemoglobin Decrease (Investigations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sensation of Foreign Body (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (N=75) | Placebo (N=75)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
Pyrexia (General disorders) | 12 (13) | 10 (10)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other